CLINICAL TRIAL: NCT06305377
Title: Turning the Tides: Achieving Rapid, Safe and Sustained Glucose Control in Adolescents With Suboptimally Controlled Type 1 Diabetes Using Advanced Hybrid Closed Loop Systems
Brief Title: Achieving Rapid, Safe and Sustained Glucose Control in Adolescents With Suboptimally Controlled Type 1 Diabetes Using Advanced Hybrid Closed Loop Systems
Status: Not yet recruiting | Type: Observational
Sponsor: Giulio Frontino (Other)
Responsible Party: Sponsor-Investigator, Giulio Frontino, sub investigator, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: DESPED-T1 study
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Tandem Control IQ — Use of Tandem control IQ in a group of diabetic adolescents in not good glicaemic control

SUMMARY:
The rational of this study is to assess if AHCL systems are able to achieve a better metabolic control (better glucometric data) after 2 weeks, 1 months. 6 months and 1 year after the start, in adolescents in not good glycaemic control.

ELIGIBILITY:
Inclusion Criteria:

* All children met the American Diabetes Association (ADA) criteria for T1D diagnosis with a current HbA1c of ≥8.5%.
* Age range 12-17 yrs old

Exclusion Criteria:

* Patients with a diagnose of genetic form of diabetes will be excluded.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: diabetics adolescents in not good glicaemic control
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-03-11 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Glucometric data | 3 months
  time in range 70-180 mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Bonfanti, MD, Principal Investigator — IRCCS San Raffaele

IPD SHARING:
Plan to Share IPD: No